CLINICAL TRIAL: NCT06625827
Title: A Study to Evaluate the Effect of Nemtabrutinib on the Pharmacokinetics of Digoxin in Healthy Participants
Brief Title: A Study of the Effect of Nemtabrutinib (MK-1026) on the Plasma Levels of Digoxin in Healthy Participants (MK-1026-012)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 1026-012; MK-1026-012 (Other: MSD)
Record Dates: First submitted 2024-10-01; First posted 2024-10-03 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2024-09

CONDITIONS: Healthy
MeSH Terms: interventions — Digoxin; ARQ531

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Digoxin (Experimental): Participants receive a single oral dose of digoxin (Treatment A).
  Interventions: Drug: Digoxin
- Digoxin + Nemtabrutinib (Experimental): Participants receive a single oral dose of digoxin coadministered with a single oral dose of nemtabrutinib (Treatment B).
  Interventions: Drug: Digoxin; Drug: Nemtabrutinib

INTERVENTIONS:
Drug: Digoxin — Oral administration
Drug: Nemtabrutinib — Oral administration
  Other Names: MK-1026; ARQ 531
  Arms: Digoxin + Nemtabrutinib

SUMMARY:
The goal of the study is to learn what happens to levels of digoxin in a healthy person's body over time. Researchers will compare what happens to digoxin in the body when it is given with and without another medicine called nemtabrutinib. Researchers are testing if digoxin levels in the body are different when digoxin is given with or without nemtabrutinib.

ELIGIBILITY:
Inclusion Criteria:

* Is in good health based on medical history, physical examination, vital signs (VS) measurements, electrocardiograms (ECGs), and laboratory safety tests performed before randomization
* Has a body mass index (BMI) 18.0 to 32.0 kg/m^2 (inclusive)

Exclusion Criteria:

* Has a medical history that may confound the results of the study or poses an additional risk to the participant in the study
* Has a hypersensitivity to digoxin and/or to other digitalis preparations including inactive ingredients (eg, lactose, corn starch and potato starch)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2023-11-07 (Actual); Primary Completion 2024-01-22 (Actual); Study Completion 2024-01-22 (Actual)

PRIMARY OUTCOMES:
Area under the Concentration-Time Curve from Time 0 to Infinity (AUC0-Inf) of Digoxin | At designated timepoints (up to approximately 7 days)
  Blood samples will be collected to determine the AUC0-Inf of digoxin.

SECONDARY OUTCOMES:
Area Under the Concentration-Time Curve from Time 0 to Last (AUC0-Last) of Digoxin | At designated timepoints (up to approximately 7 days)
  Blood samples will be collected to determine the AUC0-Last of digoxin.
Maximum Plasma Concentration (Cmax) of Digoxin | At designated timepoints (up to approximately 7 days)
  Blood samples will be collected to determine the Cmax of digoxin.
Plasma Concentration 24 Hours Postdose (C24) of Digoxin | At designated timepoints (up to approximately 24 hours)
  Blood samples will be collected to determine the C24 of digoxin.
Time to Maximum Plasma Concentration (Tmax) of Digoxin | Predose and at designated timepoints (up to approximately 7 days)
  Blood samples will be collected to determine the Tmax of digoxin.
Apparent Terminal Half-life (t1/2) of Digoxin | At designated timepoints (up to approximately 7 days)
  Blood samples will be collected to determine t1/2 of digoxin.
Apparent Clearance (CL/F) of Digoxin | At designated timepoints (up to approximately 7 days)
  Blood samples will be collected to determine the CL/F of digoxin.
Apparent Volume of Distribution (Vz/F) of Digoxin | At designated timepoints (up to approximately 7 days)
  Blood samples will be collected to determine the Vz/F of digoxin.
Number of Participants Who Experience an Adverse Event (AE) | Up to approximately 8 weeks
  An AE is any untoward medical occurrence in a participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. The number of participants who experience an AE will be reported.
Number of Participants Who Discontinue Study Due to an AE | Up to approximately 8 weeks
  An AE is any untoward medical occurrence in a participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. The number of participants who discontinue study due to an AE will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (1):
- ICON (Site 0001), Lenexa, Kansas, United States

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/